CLINICAL TRIAL: NCT05935436
Title: The Effect of Cardiac Shock Wave Therapy in the Treatment of Myocardial Infarction With Non-obstructive Coronary Arteries: a Prospective, Randomized Controlled Clinical Study
Brief Title: Cardiac Shock Wave Therapy for the Treatment of Myocardial Infarction With Non-obstructive Coronary Arteries
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ya-Wei Xu (Other)
Collaborators: Shanghai Municipal Science and Technology Commission (Other Government)
Responsible Party: Sponsor-Investigator, Ya-Wei Xu, Chief Physician, Shanghai 10th People's Hospital
Organization: Shanghai 10th People's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CSWT-MINOCA
Record Dates: First submitted 2023-06-04; First posted 2023-07-07 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Myocardial Infarction With Non-obstructive Coronary Arteries; Cardiac Shock Wave Therapy
Keywords: myocardial infarction with non-obstructive coronary arteries; cardiac shock wave therapy; D-SPECT; myocardial infarction
MeSH Terms: conditions — MINOCA; Myocardial Infarction

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CSWT Group (Active Comparator): CSWT is performed three times a week (days 1, 3, and 5) in a session with a 3-month interval between sessions or 1-month intensive treatment.
  Interventions: Device: Cardiac Shock Wave Therapy
- Control Group (Sham Comparator): Patients in the control group receive sham CSWT, the energy of cardiac shock wave therapy was the lowest, and the water bladder was in contact with the skin but not close to the skin.
  Interventions: Device: Cardiac Shock Wave Therapy

INTERVENTIONS:
Device: Cardiac Shock Wave Therapy — When operating CSWT, it is necessary to determine the target myocardium for treatment, adjust the height of the water bladder, set the energy that the patient can tolerate, and then start the treatment. During the treatment, the vital signs of the subjects should be detected.

SUMMARY:
Myocardial infarction with non-obstructive coronary arteries (MINOCA) accounts for 15% of all myocardial infarctions and its mortality rate approaches that of large vessel myocardial infarction, but there are currently no effective treatment options. Coronary microvascular dysfunction is an important mechanism of MINOCA and is closely related to adverse cardiovascular outcomes.

The prospective trial aimed to verify the safety and effectiveness of cardiac shock wave therapy (CSWT) in the treatment of Myocardial infarction with non-obstructive coronary arteries (MINOCA), and to expand the scope of clinical indications for CSWT and provide new treatment strategy for MINOCA.

DETAILED DESCRIPTION:
All participants will be fully informed of the study protocol, and informed consent will be obtained from each patient before the study. The inclusion criteria include: 1) Aged between 18 and 85 years old; 2) The initial diagnosis is acute myocardial infarction; 3) Coronary angiography shows coronary stenosis <50%; 4) Abnormal D-SPECT myocardial perfusion images; 5) Voluntary informed consent signed.

The exclusion criteria include: 1) Previous history of coronary heart disease, received percutaneous coronary intervention, coronary artery bypass surgery or myocardial infarction (MI); 2) Hemodynamic instability; 3) Acute heart failure; 4) Severe valvular heart disease requiring surgical treatment; 5) Severe liver and kidney diseases; 6) Malignant tumors with an expected survival of less than one year; 7) Patients with severe bleeding tendency; 8) Pregnant women; 9) Intervening coronary ischemic events.

Based on the literature and the number of participants with myocardial infarction in the hospital, the sample size calculated according to the formula is about 50 cases. Considering the dropout rate of 10%, the sample size should be 56 cases.

56 patients are randomly divided 1:1 by computer into the CSWT group and Control group, with 28 MINOCA participants in each group. Participants in the CSWT group are treated with conventional medical therapy (including antiplatelet drugs, statins, and antianginal drugs), combined with CSWT, and those in the Control group were treated with conventional medical therapy and sham CSWT. Care providers and physicians who follow participants (parameters of this study) should be blinded to group assignment. CSWT is performed according to the recommended protocol on shock wave output and the number of shots delivered per point developed by Tohoku University, Japan, and with protocol equipment (Modulith SLC; Storz Medical, Switzerland) developed by the University of Essen, Germany. CSWT is performed three times a week (days 1, 3, and 5) in a session with a 3-month interval between sessions or 1-month intensive treatment. 40 The participants underwent CSWT for 3 months and 9 CSWT sessions were performed in total. Participants in the control group received sham CSWT, the energy of cardiac shock wave therapy was the lowest, and the water bladder was in contact with the skin but not close to the skin.

Examinations in this prospective trial include D-SPECT, blood biochemical examination, myocardial marker, and cardiopulmonary exercise testing. During follow-up, investigators will record major adverse cardiovascular events, and adverse events caused by other treatments. The safety and effectivity of CSWT will be verified by clinical parameters, D-SPECT, and peak oxygen consumption in CPET.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 85 years old
* The initial diagnosis is acute myocardial infarction
* Coronary angiography shows coronary stenosis <50%
* Abnormal D-SPECT myocardial perfusion images
* Voluntary informed consent signed

Exclusion Criteria:

* Previous history of coronary heart disease, received percutaneous coronary intervention, coronary artery bypass surgery or myocardial infarction (MI)
* Hemodynamic instability
* Acute heart failure
* Severe valvular heart disease requiring surgical treatment
* Severe liver and kidney diseases
* Malignant tumors with expected survival of less than one year
* Patients with severe bleeding tendency
* Pregnant women
* Intervening coronary ischemic events

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-06-20 (Estimated)

PRIMARY OUTCOMES:
Change from baseline myocardial infarct area at 6 months | 1 day of inclusions and 6 months after the first treatment.
  The location and extent of myocardial infarction were determined by D-SPECT.

SECONDARY OUTCOMES:
Change from baseline peak oxygen consumption at 6 months | 1 day of inclusions and 6 months after the first treatment.
  maximum kilogram oxygen uptake accessed during Cardiopulmonary Exercise Testing (CPET)
Change from baseline myocardial marker at 6 months | 1 day of inclusions and 6 months after the first treatment.
  creatine kinase phosphate-isozyme (CK-MB) in blood samples
Change from baseline hepatorenal function indexes at 6 months | 1 day of inclusions and 6 months after the first treatment.
  alanine aminotransferase (ALT), aspartate aminotransferase (AST), and serum creatinine (SCr) in blood samples

OTHER OUTCOMES:
Major adverse cardiovascular events (MACE) | From the date of inclusion until the date of documented adverse events with 6 months
  cardiovascular death, non-fatal myocardial infarction, unplanned coronary revascularization, stroke, heart failure, and angina-related rehospitalization
Other treatment-related adverse reactions | From the date of inclusion until the date of treatment-related adverse reactions within 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Cardiology, Shanghai Tenth People's Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes